CLINICAL TRIAL: NCT05428046
Title: Preventing Eating Disorders by Improving Mental Health Literacy in Chinese Adolescents: A Non-randomized Cluster Controlled Trial
Brief Title: Preventing Eating Disorders by Improving Mental Health Literacy in Chinese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHL-ED
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Eating Disorders; Mental Health Literacy
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHL intervention (Experimental): Mental health literacy intervention for eating disorder
  Interventions: Behavioral: MHL intervention
- Waiting list (Other): The waiting list group received MHL intervention at the end of 12 weeks follow-up assessment.
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: MHL intervention — The current MHL intervention is a brief online intervention and comprises two modules. The first module is a short video introducing a teenage girl with bulimia nervosa. The second module is an online lecture comprising information about eating disorders including the prevalence, symptoms, type, cause, treatment, a related symptom checker, and sources of help. The above two modules are implemented in a single session lasting approximately 2 hours.
  Arms: MHL intervention
Behavioral: Waiting list — Participants assigned to the waiting list group will not receive any intervention until the end of the 12 weeks follow-up. They received the same intervention as the MHL intervention group after the 12 weeks follow-up test.
  Arms: Waiting list

SUMMARY:
Mental health literacy (MHL) is necessary for the prevention, detection, and treatment of eating disorders, whereas the MHL about eating disorders is inadequate in China. Thus, the current study aimed to improve the MHL for eating disorders among Chinese adolescents via a brief online intervention.

ELIGIBILITY:
Inclusion Criteria:

* Middle school students

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Eating disorders mental health literacy | pre-intervention, post-intervention, 4 weeks follow-up, 12 weeks follow-up
  The vignette for eating disorders mental health literacy was developed for the current study. The vignette describes a 14-year old girl who has bulimia nervosa. We also conducted a 5-point Likert scale to assess the knowledge, attitude, and help-seeking behaviors of eating disorders. Higer scores indicating a higer level of eating disorders mental health literacy.
social distance scale | pre-intervention, post-intervention, 4 weeks follow-up, 12 weeks follow-up
  The social distance scale was used to assess the level of social rejection that participants were likely to impose on people with eating disorders. The lower the score, the greater the desire for social distancing and the more negative the attitude toward people with eating disorders.

SECONDARY OUTCOMES:
Weight Concerns Scale | pre-intervention, post-intervention, 4 weeks follow-up, 12 weeks follow-up
  The Weight Concerns Scale was used to assess weight concern and shape concern, with a higher score indicating more concerns.
The SCOFF | pre-intervention, post-intervention, 4 weeks follow-up, 12 weeks follow-up
  The SCOFF (Sick, Control, One, Fat, Food) was used to detect the existence of eating disorder symptoms. Scores of 2 or greater were originally set a cut-off point for maximum sensitivity to detect anorexia and Bulimia nervosa (Morgan et al, 1999).
Actual help-seeking behavior | pre-intervention, post-intervention, 4 weeks follow-up, 12 weeks follow-up
  We conducetd three items to assess the actual help-seeking behavior, including, "In the last 6 months, have you come into contact with someone who you think may have the same problems as Lily?","Have you offered help to them?", "How you helped him/her?".
Patient Health Questionnaire-4 | pre-intervention, post-intervention, 4 weeks follow-up, 12 weeks follow-up
  The Patient Health Questionnaire-4 was used to assess any negative impact on participant's well-being. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided